CLINICAL TRIAL: NCT00187707
Title: Influence of Intestinal Transporter Genetic Variants on the Bioavailability of Gabapentin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1003
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gabapentin (Other): Subjects will take a single dose of 400 mg of gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Subjects will take a single dose of 400 mg of gabapentin
  Other Names: NEURONTIN

SUMMARY:
The current study is part of a large multi-investigator grant to look at the pharmacogenetics of a number of membrane transporters. Previously, we have recruited a cohort of healthy volunteers (Studies of Pharmacogenetics in Ethnically-diverse Populations, or SOPHIE) and have resequenced the coding region of a number of membrane transporter genes to identify genetic polymorphisms in these genes. We plan to take a genotype-to-phenotype approach to study the influence of specific polymorphisms in the intestinal transporters, such as the novel organic cation transporters 1 and 2 (OCTN1 and OCTN2) genes on the bioavailability of gabapentin in healthy subjects. Eligible subjects will have a single inpatient study visit, during which they will take a single dose of gabapentin, and provide blood and urine samples over the course of 36 hours (5 terminal elimination gabapentin half-lives) for pharmacokinetic analysis.

DETAILED DESCRIPTION:
Detailed description pending

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have previously participated in the "SOPHIE" study.
* Subjects will be between the ages of 18 and 40 years old
* Subjects will have been selected as healthy by medical history questionnaire and screening blood work (CBC, Comprehensive Metabolic panel).
* Subjects will be taking no regular medications and will have normal renal function.

Exclusion Criteria:

* Pregnant
* Have a new history indicating they are no longer healthy; Individuals with anemia (hemoglobin < 12 g/dL), an elevation in liver enzymes to higher than double the respective normal value, or elevated creatinine concentrations (males ≥ 1.5 mg/dL, females ≥ 1.4 mg/dL), will be excluded.
* Taking a medication that could confound study results
* Do not consent to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Influence of Intestinal Transporter Genetic Variants on the Bioavailability of Gabapentin | Gabapentin
  To evaluate the bioavailability of Gabapentin in healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States